CLINICAL TRIAL: NCT03142009
Title: Family Listening Program: Multi-Tribal Implementation and Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-289
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Substance Abuse
Keywords: Community-Based Participatory Research
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The investigators use a two arm non-equivalent control group design with pretest, immediate post- test, and 12 month follow-up assessment points. Among quasi-experimental designs that could be employed, this design carries several advantages over other designs in being able to infer causality. One advantage of this design is that it allows for a more meaningful analysis of the impact of the FL/CP intervention by a comparison of the intervention group with the usual and customary comparison group, an advantage not possible with single-group over time designs. Second, the design provides an analysis of diffusion effects (i.e. the potential influence of the intervention on the comparison group over time). Given the tight social networks and small number of interconnected families in the three participating communities, the investigators expect some degree of program diffusion in the comparison group families.
Masking Description: Due to factors that make the randomization of participants to either an intervention or usual and customary treatment group not feasible, the investigators do not use randomization or masking. Only children's data are analyzed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program group (Experimental): Tribal Research Team members recruit participants by sending letters home with the fourth and fifth grade children. This letter provides an overview of the FL/CP and invite interested parents and children to learn more. TRT and UNM team members follow-up with interested parents individually. If families are committed to being a part of FL/CP, a meeting is set to conduct the informed consent process and complete pretest. Families in the program group then attend FL/CP sessions which covers the intergenerational culturally adapted curriculum. Program families also participate in various aspects of the program including completing a Community Action Project.
  Interventions: Other: Intergenerational culturally adapted curriculum
- Comparison group (No Intervention): Upon receiving the letter families that selected not to participate or who decline to participate will be invited to take part in the research study as comparison participants. Comparison participants do not attend the FL/CP sessions and only complete the pre, post and 1 year post tests.

INTERVENTIONS:
Other: Intergenerational culturally adapted curriculum — Each session starts with a collective dinner with families eating together. Then practice their Indian and clan names. The sessions are led by facilitators in their own language or bilingually. The facilitators then divide the families into children and adult groups to address the theme of the session, and they then return together at the end of the session to share their learnings. The sessions always end with the children and adults writing in their journals which are individual pages that they then put in their curriculum binders. Families are then given their "home practice," which is a task that the families do together during the intervening week. The facilitators collect the curriculum binders after each session to bring back to the families the next week.
  Arms: Program group

SUMMARY:
This is a five-year R01 effectiveness trial where tribal partners are committed to assessing the Family Listening/Circle Program's effectiveness and disseminating the approach and intervention within Indian Country as a best practice in reducing substance abuse health disparities.Three specific aims of the grant are 1) To rigorously test effectiveness of FLCP; with a comparative longitudinal design within and across the tribes, with 4th graders to prevent substance initiation/use and strengthen families; 2) Through CBPR, support TRTs to transform their research capacities into local prevention research infrastructures and partnering; 3)To assess additional program effects on other health/education programs and leadership within the tribes. In sum, this multi-tribal/academic partnership builds on accomplishments to test the effectiveness of an innovative intervention. This grant provides an unparalleled opportunity to reduce substance abuse in three tribal communities, strengthen tribal research capacities, and impact substance abuse prevention research designs nationally, by illustrating how CBPR processes can integrate evidence-based and cultural-centered practices to create effective programs that generate community ownership and sustainability.

DETAILED DESCRIPTION:
With substance abuse concerns plaguing tribal communities, health preventive approaches for American Indian (AI) children need urgent attention. Mainstream programs fall short by failing to speak to AI children on their own terms. Not so with the Family Listening/Circle Program (FL/CP) which integrates an evidence-based family-strengthening core, with cultural values and practices for 4th graders, their parents and elders. Through previous Native American Research Centers for Health funding (Indian Health Service & National Institutes of Health partnership) the FL/CP was created and piloted by community-based participatory research (CBPR) partnerships between the University of New Mexico Center for Participatory Research and three tribal communities: Pueblo of Jemez, Ramah Band of Navajo and Mescalero Apache Nation. FL/CP fills a gap in substance abuse prevention by recapturing historic traditions of cultural transmission, such as family dinner story-telling where elders connect with children, supporting enhanced child-family communication and psycho-social coping through traditional dialogue, indigenous languages and empowerment where children and families create community action projects addressing community substance abuse. With initial FL/CP pilot and feasibility research completed, Tribal Research Teams (TRTs) from the Pueblo of Jemez, Ramah Band of Navajo and Mescalero Apache Nation are now in place for full program implementation and effectiveness testing through a longitudinal quasi-experimental design involving a long-term, multi-tribal/academic research partnership. Under this five-year R01 effectiveness trial, tribal partners are committed to assessing the program's effectiveness and disseminating the approach and intervention within Indian Country as a best practice in reducing substance abuse health disparities, with TRTs collaborating on all research activities, implementation, interpretation/analysis, and dissemination plans. Three specific aims are 1) To rigorously test effectiveness of FLCP; with a comparative longitudinal design within and across the tribes, with 4th graders to prevent substance initiation/use and strengthen families; 2) Through CBPR, support TRTs to transform their research capacities into local prevention research infrastructures and partnering; 3)To assess additional program effects on other health/education programs and leadership within the tribes. In sum, this multi-tribal/academic partnership builds on accomplishments to test the effectiveness of an innovative intervention. This grant provides an unparalleled opportunity to reduce substance abuse in three tribal communities, strengthen tribal research capacities, and impact substance abuse prevention research designs nationally, by illustrating how CBPR processes can integrate evidence-based and cultural-centered practices to create effective programs that generate community ownership and sustainability.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria includes any families from Mescalero Apache, Jemez Pueblo and Ramah Navajo with a fourth and fifth-grade child and their parents or guardian, and grandparents who will volunteer to participate. Only children's data are analyzed.

-

Exclusion Criteria:Those whom are ineligible in this study are: those that do not give consent and/or assent to participate; those that do not identify as tribal members of Mescalero Apache, Jemez Pueblo and Ramah Navajo or as the family member of someone that identifies as Mescalero Apache, Jemez Pueblo and Ramah Navajo; children and that are not in the targeted range of fourth and fifth grade.

-

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 266 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenda Belone, PhD, Principal Investigator — University of New Mexico; Nina Wallerstein, DrPH, Principal Investigator — University of New Mexico
Locations (3):
- United States (3):
  - Pueblo of Jemez Department of Education, Jemez Pueblo, New Mexico
  - Mescalero Prevention Program, Mescalero, New Mexico
  - Ramah Navajo School Board, Pinehill, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallerstein N, Duran B. Community-based participatory research contributions to intervention research: the intersection of science and practice to improve health equity. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S40-6. doi: 10.2105/AJPH.2009.184036. Epub 2010 Feb 10. PMID 20147663
- [Background] Beauvais F. An integrated model for prevention and treatment of drug abuse among American Indian youth. J Addict Dis. 1992;11(3):63-80. doi: 10.1300/J069v11n03_04. PMID 1627667
- [Background] Mail PD, Johnson S. Boozing, sniffing, and toking: an overview of the past, present, and future of substance use by American Indians. Am Indian Alsk Nativ Ment Health Res (1987). 1993;5(2):1-33. doi: 10.5820/aian.0502.1993.1. PMID 8130311
- [Background] Beauvais F. Preventing Drug Abuse among Native American Young People. 1980, Fort Collins, CO: Western Behavioral Studies.
- [Background] Beauvais F. Preventing Drug Abuse among Native American Young People. 1996, Ft. Collins, CO: Western Behavioral Studies
- [Background] Okwumabua JO, Duryea EJ. Age of onset, periods of risk, and patterns of progression in drug use among American Indian high school students. Int J Addict. 1987 Dec;22(12):1269-76. doi: 10.3109/10826088709027486. PMID 3436694
- [Background] Swaim RC, Oetting ER, Edwards RW, Beauvais F. Links from emotional distress to adolescent drug use: a path model. J Consult Clin Psychol. 1989 Apr;57(2):227-31. doi: 10.1037//0022-006x.57.2.227. PMID 2708609
- [Background] NMDOH, Racial and ethnic health disparities report card, O.o.P.a.M. Health, Editor, 2007, NMDOH: Department of Health Santa Fe, NM. p. 1-24.
- [Background] Szlemko WJ, Wood JW, Thurman PJ. Native Americans and alcohol: past, present, and future. J Gen Psychol. 2006 Oct;133(4):435-51. doi: 10.3200/GENP.133.4.435-451. PMID 17128961
- [Background] Miller WR. Motivational interviewing: research, practice, and puzzles. Addict Behav. 1996 Nov-Dec;21(6):835-42. doi: 10.1016/0306-4603(96)00044-5. PMID 8904947
- [Background] Borowsky IW, Resnick MD, Ireland M, Blum RW. Suicide attempts among American Indian and Alaska Native youth: risk and protective factors. Arch Pediatr Adolesc Med. 1999 Jun;153(6):573-80. doi: 10.1001/archpedi.153.6.573. PMID 10357296
- [Background] United States Census, B., 2010 Census Interactive Population Search: New Mexico, 2010.
- [Background] Racial and Ethnic Health Disparities Report Card, 7th Edition, N.M.D.o. Health, Editor 2012, Office of Health Equity, Office of Policy and Accountability: Santa Fe, NM. p. 1-43.
- [Background] New Mexico Youth Risk and Resiliency Survey (YRRS): American Indian High School Students - Aggregate Report, 2009, New Mexico Department of Health, New Mexico Public Education Department, University of New Mexico Prevention Research Center, Albuquerque Area Southwest Tribal Epidemiology Center. p. 1-197.
- [Background] Oetting ER, Swaim RC, Edwards RW, Beauvais F. Indian and Anglo adolescent alcohol use and emotional distress: path models. Am J Drug Alcohol Abuse. 1989;15(2):153-72. doi: 10.3109/00952998909092718. PMID 2729224
- [Background] Conger RD. The social context of substance abuse: a developmental perspective. NIDA Res Monogr. 1997;168:6-36. No abstract available. PMID 9260163
- [Background] Conger RD, Lorenz FO, Elder GH, Melby JN, Simons RL, Conger KJ. A process model of family economic pressure and early adolescent alcohol use. The Journal of Early Adolescence 11(4): 430, 1991
- [Background] Loeber, R. Antisocial behavior and mental health problems explanatory factors in childhood and adolescence. 1998; Available from: http://search.ebscohost.com/login.aspx?direct=true&scope=site&db=nlebk&db=nlabk&AN=19368.
- [Background] Gottesman IL, Goldsmith HH. Developmental Psychology of Antisocial Behaviors: Interting Genes into its Ontogenesis and Epigenesis, in Threats to Optimal Development: Integrating Biological, Psychological and Social Risk Factors, C.A. Nelson, Editor. 1994
- [Background] Lahey BB, Piacentini JC, McBurnett K, Stone P, Hartdagen S, Hynd G. Psychopathology in the parents of children with conduct disorder and hyperactivity. J Am Acad Child Adolesc Psychiatry. 1988 Mar;27(2):163-70. doi: 10.1097/00004583-198803000-00005. No abstract available. PMID 3360717
- [Background] O'Connor TG, McGuire S, Reiss D, Hetherington EM, Plomin R. Co-occurrence of depressive symptoms and antisocial behavior in adolescence: a common genetic liability. J Abnorm Psychol. 1998 Feb;107(1):27-37. doi: 10.1037//0021-843x.107.1.27. PMID 9505036
- [Background] Silberg J, Rutter M, Meyer J, Maes H, Hewitt J, Simonoff E, Pickles A, Loeber R, Eaves L. Genetic and environmental influences on the covariation between hyperactivity and conduct disturbance in juvenile twins. J Child Psychol Psychiatry. 1996 Oct;37(7):803-16. doi: 10.1111/j.1469-7610.1996.tb01476.x. PMID 8923223
- [Background] Duran B. Duran E, Braveheart MYH. Native Americans and the trauma of history, in Studying Native America: Problems and Prospects in Native American Studies, R. Thornton, Editor. 1998, University of Wisconsin Press: Madison.
- [Background] Duran E, Duran B. Native American postcolonial psychology. 1995, Albany, NY US: State University of New York Press.
- [Background] Duncan TE, Tildesley E, Duncan SC, Hops H. The consistency of family and peer influences on the development of substance use in adolescence. Addiction. 1995 Dec;90(12):1647-60. doi: 10.1046/j.1360-0443.1995.901216477.x. PMID 8555956
- [Background] Dinges MM, Oetting ER. Similarity in drug use patterns between adolescents and their friends. Adolescence. 1993 Summer;28(110):253-66. PMID 8317274
- [Background] Hawkins EH, Cummins LH, Marlatt GA. Preventing substance abuse in American Indian and Alaska native youth: promising strategies for healthier communities. Psychol Bull. 2004 Mar;130(2):304-23. doi: 10.1037/0033-2909.130.2.304. PMID 14979774
- [Background] Kandel DB, Yamaguchi K, Chen K. Stages of progression in drug involvement from adolescence to adulthood: further evidence for the gateway theory. J Stud Alcohol. 1992 Sep;53(5):447-57. doi: 10.15288/jsa.1992.53.447. PMID 1405637
- [Background] Rutter M. Psychosocial resilience and protective mechanisms. Am J Orthopsychiatry. 1987 Jul;57(3):316-331. doi: 10.1111/j.1939-0025.1987.tb03541.x. PMID 3303954
- [Background] Catalano RF, Berglund ML, Ryan JAM, Lonczak HS, Hawkins JD. Positive Youth Development in the United States: Research Findings on Evalutions of Positive Youth Development Programs. Annals of the American Academy of Political and Social Science, 2004. 591(1): p. 98.
- [Background] Kumpfer KL, Molgaard V, Spoth R. The Strengthening Families Program for the prevention of delinquency and drug use, R.D. Peters and R.J. McMahon, Editors. 1996, Sage Publications Inc: Thousand Oaks, CA US. p. 241.
- [Background] Brody GH, Chen YF, Kogan SM, Yu T, Molgaard VK, DiClemente RJ, Wingood GM. Family-centered program deters substance use, conduct problems, and depressive symptoms in black adolescents. Pediatrics. 2012 Jan;129(1):108-15. doi: 10.1542/peds.2011-0623. Epub 2011 Dec 12. PMID 22157131
- [Background] Whitbeck LB, Hoyt Dr, Stubben JD, LaFromboise T. Traditional culture and academic success among American Indian children in the upper Midwest. Journal of American Indian Education 40(2): 48, 2001
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Dumont M, Provost MA. Resilience in adolescents: Protective role of social support, coping strategies, self-esteem, and social activities on experience of stress and depression. Journal of Youth and Adolescence 28(3): 343, 1999
- [Background] Whitbeck LB, McMorris BJ, Hoyt DR, Stubben JD, Lafromboise T. Perceived discrimination, traditional practices, and depressive symptoms among American Indians in the upper midwest. J Health Soc Behav. 2002 Dec;43(4):400-18. PMID 12664673
- [Background] Whitbeck LB, Hoyt DR, McMorris BJ, Chen X, Stubben JD. Perceived discrimination and early substance abuse among American Indian children. J Health Soc Behav. 2001 Dec;42(4):405-24. PMID 11831140
- [Background] Coggins K, Williams E, Radin N. The Traditional Values of the Ojibwe Parents and the School Performance of their Children: An Exploratory Study. Journal of American Indian Education 36(3): 1, 1997
- [Background] Pankratz MM, Jackson-Newsom J, Giles SM, Ringwalt CL, Bliss K, Bell ML. Implementation fidelity in a teacher-led alcohol use prevention curriculum. J Drug Educ. 2006;36(4):317-33. doi: 10.2190/H210-2N47-5X5T-21U4. PMID 17533804
- [Background] Cajete G. Look to the Mountain: An Ecology of Indigenous Education. First Edition. 1994: Kivaki Press 585 E. 31st St. Durango CO 81301
- [Background] Wallerstein, N., Evidence of effectiveness of empowerment interventions to reduce health disparities and social exclusion. Health Evidence Network, 2006.
- [Background] Altman DG, Feighery EC. Future directions for youth empowerment: commentary on application of youth empowerment theory to tobacco control. Health Educ Behav. 2004 Oct;31(5):641-7. doi: 10.1177/1090198104268683. No abstract available. PMID 15358895
- [Background] Holden DJ, Messeri P, Evans WD, Crankshaw E, Ben-Davies M. Conceptualizing youth empowerment within tobacco control. Health Educ Behav. 2004 Oct;31(5):548-63. doi: 10.1177/1090198104268545. PMID 15358889
- [Background] Berg M, Coman E, Schensul JJ. Youth Action Research for Prevention: a multi-level intervention designed to increase efficacy and empowerment among urban youth. Am J Community Psychol. 2009 Jun;43(3-4):345-59. doi: 10.1007/s10464-009-9231-2. PMID 19387823
- [Background] Lipari L. Listening, Thinking, Being. Communication Theory. 20(3): 348, 2010
- [Background] Wallerstein N, Auerbach E. Problem-posing at work: Popular educator's guide. 2004: Grass Roots Press.
- [Background] Pueblo of Jemez. [cited 2013 April 27]; Available from: http://www.jemezpueblo.org/.
- [Background] Wallerstein N, Duran BM, Aguilar J, Joe L, Loretto F, Toya A, Yepa-Waquie H, Padilla R, Shendo K. Jemez Pueblo: built and social-cultural environments and health within a rural American Indian community in the Southwest. Am J Public Health. 2003 Sep;93(9):1517-8. doi: 10.2105/ajph.93.9.1517. No abstract available. PMID 12948972
- [Background] English KC, Wallerstein N, Chino M, Finster CE, Rafelito A, Adeky S, Kennedy M. Intermediate outcomes of a tribal community public health infrastructure assessment. Ethn Dis. 2004 Summer;14(3 Suppl 1):S61-9. PMID 15682773
- [Background] Cashman SB, Adeky S, Allen AJ 3rd, Corburn J, Israel BA, Montano J, Rafelito A, Rhodes SD, Swanston S, Wallerstein N, Eng E. The power and the promise: working with communities to analyze data, interpret findings, and get to outcomes. Am J Public Health. 2008 Aug;98(8):1407-17. doi: 10.2105/AJPH.2007.113571. Epub 2008 Jun 12. PMID 18556617
- [Background] Oetzel J, Wallerstein N, Solimon A, Garcia B, Siemon M, Adeky S, Apachito G, Caston E, Finster C, Belone L, Tafoya G. Creating an instrument to measure people's perception of community capacity in American Indian communities. Health Educ Behav. 2011 Jun;38(3):301-10. doi: 10.1177/1090198110379571. Epub 2011 Apr 5. PMID 21467256
- [Background] Spoth R, Redmond C. Illustrating a Framework for Rural Prevention Research: Project Family Studies of Rural Families Participation and Outcomes, in Preventing Childhood Disorders, Substance Abuse, and Delinquency, R.D. Petters and R.J. McMahon, Editors. 1996, Sage Publications: Thousand Oaks, CA.
- [Background] Spoth R, Redmond C, Haggerty K, Ward T. A Controlled Parenting Skills Outcome Study Examining Individual Difference and Attendance Effects. Journal of Marriage & Family 57(2): 449, 1995.
- [Background] Whitbeck, L.B., Bii-zin-da-de-da: The listening to one another prevention program. Workshop presented at the Second National Conference on Drug Abuse Prevention Research: A Progress Update, Washington, DC, 2001.
- [Background] Dutta A. Development-induced displacement and human rights. 2007, New Dilhi: Deep & Deep Publications.
- [Background] Hall GC. Psychotherapy research with ethnic minorities: empirical, ethical, and conceptual issues. J Consult Clin Psychol. 2001 Jun;69(3):502-10. doi: 10.1037//0022-006x.69.3.502. PMID 11495179
- [Background] Hawe P, Shiell A, Riley T. Theorising interventions as events in systems. Am J Community Psychol. 2009 Jun;43(3-4):267-76. doi: 10.1007/s10464-009-9229-9. PMID 19390961
- [Background] Wang CC. Youth participation in photovoice as a strategy for community change. Journal of Community Practice 14(1): 147, 2006
- [Background] Dutta MJ. Communicating about culture and health: Theorizing culture-centered and cultural sensitivity approaches. Communication Theory 17(3): 304, 2007
- [Background] World Health, O. Committee on Indigenous Health. (1999, 2007). The Geneva Declaration on the Health and Survival of Indigenous Peoples (WHO/HSD/00.1.). United Nations Declaration on the Rights of Indigenous Peoples, adopted by General Assembly, 2007 (A/RES/61/295). [cited 2011 01/17]; Available from: http://www.un.org/esa/socdev/unpfii/en/declaration.html.
- [Background] Shendo K, Toya A, Tafoya E, Yepa M, Tosa J, Yepa T, Yepa-Waquie H, Gachupin D, Gachupin C, Yepa K, Rae R, Belone L, Tafoya G, Noyes E, Wallerstein N. An Intergenerational Family Community-Based Participatory Research Prevention Program: Hemish of Walatowa Family Circle Program. IHS Prim Care Provid. 2012 Aug;37(8):185-191. No abstract available. PMID 35498637
- [Background] Belone L. et al/ Using participatory research to address substance use in an American-Indian community, in Communication Activism: Struggling for social justice amidst difference, L.R. Frey and K.M. Carragee, Editors. Hampton Press, Inc.: New York, NY. p. 403-434, 2012
- [Background] Israel BA, Schulz AJ, Parker EA, Becker AB. Review of community-based research: assessing partnership approaches to improve public health. Annu Rev Public Health. 1998;19:173-202. doi: 10.1146/annurev.publhealth.19.1.173. PMID 9611617
- [Background] Israel BA., et al., eds. Methods In CBPR for Health. 2nd ed. Jossy-Bass: San Francisco, 2012
- [Background] Walters KL, et al., 'Indigenist' collaborative research efforts in Native American communities, A.R. Stiffman, Editor. Oxford University Press: New York, NY US. p. 146, 2009
- [Background] Laveaux D, Christopher S. Contextualizing CBPR: Key Principles of CBPR meet the Indigenous research context. Pimatisiwin. 2009 Jun 1;7(1):1. PMID 20150951
- [Background] Minkler M, Wallerstein N. Community-Based Participatory Research for Health: From Process to Outcomes. 2nd ed. Jossey-Bass: San Francisco, 2008
- [Background] Brownson RC, Colditz GA, Proctor EK. Dissemination and implementation research in health : translating science to practice. 2012: Oxford ; New York : Oxford University Press 2012.
- [Background] Cook TD, Campbell DT. Quasi-Experimentation: Design & Analysis Issues for Field Settings. Boston: Houghton-Mifflin, 1979.
- [Background] Buchanan DR, Miller FG, Wallerstein N. Ethical issues in community-based participatory research: balancing rigorous research with community participation in community intervention studies. Prog Community Health Partnersh. 2007 Summer;1(2):153-60. doi: 10.1353/cpr.2007.0006. PMID 20208234
- [Background] Hicks S, Duran B, Wallerstein N, Avila M, Belone L, Lucero J, Magarati M, Mainer E, Martin D, Muhammad M, Oetzel J, Pearson C, Sahota P, Simonds V, Sussman A, Tafoya G, Hat EW. Evaluating community-based participatory research to improve community-partnered science and community health. Prog Community Health Partnersh. 2012 Fall;6(3):289-99. doi: 10.1353/cpr.2012.0049. PMID 22982842
- [Background] Pearson C., et al., CBPR Variable Matrix: Research for Improved Health in Academic-Community Partnerships.CES4Health.info. 2011.
- [Background] Garcia LF, Aluja A, Del Barrio V. Testing the hierarchical structure of the Children's Depression Inventory: a multigroup analysis. Assessment. 2008 Jun;15(2):153-64. doi: 10.1177/1073191107310310. PMID 18463406
- [Background] Greenspoon PJ, Saklofske DH. Validity and reliability of the multidimensional student's life satisfaction scale with Canadian children. Journal of psychoeducational assessment 15: 138-155, 1997.
- [Background] Hanson TL, Kim JO. Measuring resilience and youth development: the psychometric properties of the health Kids Survey. Wahington, DC: U.S. Department of Education, Institute of Education Sciences, National Center for Education Evaluation and Regional Assistance, Regional Educational Laboratory West Retrieved from http://ies.ed.gov/ncee/edlabs. 2007
- [Background] Kovacs M. Children's Depression Inventory. New York, NY: Multi-Health Systems, 1992.
- [Background] March JS, Parker JD, Sullivan K, Stallings P, Conners CK. The Multidimensional Anxiety Scale for Children (MASC): factor structure, reliability, and validity. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):554-65. doi: 10.1097/00004583-199704000-00019. PMID 9100431
- [Background] Orvaschel H, Weissman MM, Padian N, Lowe TL. Assessing psychopathology in children of psychiatrically disturbed parents: A pilot study. J Am Acad Child Psychiatry. 1981 Winter;20(1):112-22. doi: 10.1016/s0002-7138(09)60721-4. No abstract available. PMID 7217544
- [Background] Weissman MM, Orvaschel H, Padian N. Children's symptom and social functioning self-report scales. Comparison of mothers' and children's reports. J Nerv Ment Dis. 1980 Dec;168(12):736-40. doi: 10.1097/00005053-198012000-00005. PMID 7452212
- [Background] Wilson N, Minkler M, Dasho S, Wallerstein N, Martin AC. Getting to social action: the Youth Empowerment Strategies (YES!) project. Health Promot Pract. 2008 Oct;9(4):395-403. doi: 10.1177/1524839906289072. Epub 2006 Jun 27. PMID 16803932
- [Background] Zimmerman, M. Empowerment Theory: Psychological, Organizational and Community Levels of Analysis. In J. Rappaport (Ed.), Handbook of Community Psychology. New York: Kluwer Academic/Plenum Publishing, 2000.
- [Background] Zimmerman MA, Ramirez-Valles J, Washienko KM, Walter B, Dyer S. The development of a measure of enculturation for Native American youth. Am J Community Psychol. 1996 Apr;24(2):295-310. doi: 10.1007/BF02510403. PMID 8795263
- [Background] Belone L, Tosa J, Shendo K, Toya A, Straits K, Tafoya G, Rae R, Noyes E, Bird D, Wallerstein N. Community Based Participatory Research for Cocreating interventions with Native communities: a partnership between the University of New Mexico and The Pueblo of Jemez. In Zane N, Bernal G, Leong FTL, ed. Evidence Based Psychological Practices With Ethnic Minorities. American Psychological Association (APA); 2016: 199-220.
- [Background] Belone L, Oetzel JG, Wallerstein N, Tafoya G, Rae R, Rafelito A, Kelhoyouma L, Burbank I, Finster C, Henio-Charley J, Maria PG, Thomas A. Using participatory research to address substance use in an American-Indian community. In Frey LR, Carragee KM, ed. Communication Activism: Struggling for social justice amidst difference. New York, NY: Hampton Press, Inc; 2012: 403-434.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of children participants occurred in three tribal communities: Ramah Navajo, Mescalero Apache Tribe, and Pueblo of Jemez. UNM Health Sciences Human Research Protections Office (HRPO) approved recruitment from 2014 for up to 12 families (typically one child and one caregiver) from each tribal community for the full five years of the study, with the official closing of the IRB on Feb 6, 2021. Tribes recruited students from different schools in their communities. Parents not analyzed
Period: Overall Study
Arm/Group | Program Group | Comparison Group
Started | 138 (Children were recruited from the fourth and fifth grades and later extended with NIH approval to the sixth grade to take pre and post-tests and one year follow-up post-tests. We analyzed by post test and one-year post. Data reported is by one year post. Their parents were also recruited to take pre and post-tests. The numbers in this report represent the children (as there is only one place to put the numbers of participants). Interviews were also collected from tribal program staff.) | 128 (Children were recruited from the same grades as the intervention children and, if their families chose not to participate, were placed in the comparison group to take pre and post-tests. Their parents were also recruited to take pre and post-tests and one year follow-up post-tests. We analyzed by post test and one-year post. Data reported is by one year post. The numbers in this report represent the children (as there is only one place to put the numbers of participants).)
Completed | 93 (All tribes completed recruitment) | 98 (All tribes completed recruitment)
Not Completed | 45 | 30
Not completed — Lost to Follow-up | 45 | 30

BASELINE CHARACTERISTICS:
Population: No difference from assignment in participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Program Group | Comparison Group | Total
Number analyzed (Participants) | 138 | 128 | 266
Age, Continuous [Mean (Full Range); unit: years] | 10 [8 to 12] | 10 [9 to 12] | 10 [8 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 69 | 140
  Male | 67 | 59 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Tribal members | 138 | 128 | 266
Region of Enrollment [Number; unit: participants]
  United States | 138 | 128 | 266
Depression [Mean (Standard Deviation); unit: units on a scale] — Depression scale (validated for children) items were coded 1 to 3, and the arithmetic mean of 26 items was used to compute the scale. The scale has a minimum of 1.0 and a maximum of 3.0 with higher values be better, i.e. lower levels of depression. Children took pre-test survey, post-test (2-4 months after intervention), and one year post after the intervention.
  units on a scale | 2.63 (0.25) | 2.71 (0.23) | 2.67 (0.24)

OUTCOME MEASURES:

1. Primary Outcome: Child Well-being
Description: Self-report measures of anxiety, Anxiety Panic/GAD Sub-Scale, average change from baseline (pre-program participation). Anxiety Items coded are coded 1-4. The scale was calculated as the arithmetic average of items, which results in a minimum value of 1 and a maximum value of 4. Lower scores are better. The Panic/GAD sub-scale was the average of three items with the same min/max as the full scale. Children surveyed at pre-test, post-test (2-4 months after intervention), and one-year post intervention.
Time Frame: post-test (2-4 months after intervention)
Population: Children age 10-12 recruited from three different tribal communities, with program families recruited from children in schools, with program families agreeing to participate and families who did not participate allocated to comparison group. 4 intervention children and 2 comparison children did not complete post-survey (2-4 months). Because this average looks at the difference in mean change between two arms, therefore negative means are possible. This represents a change that is favorable.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Program Group | Comparison Group
Number analyzed (Participants) | 134 | 126
units on a scale | -0.20 [-0.34 to -0.05] | 0.05 [-0.10 to 0.20]
Statistical Analysis 1: Comparison: Program Group vs Comparison Group; Test type: Superiority; p = .021, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-.45 to -.04]

2. Secondary Outcome: Child Well-being
Description: Self-report measures of depression, change from baseline at one-year, Depression scale items were coded 1 to 3, and the arithmetic mean of 26 items was used to compute the scale. The scale has a minimum of 1.0 and a maximum of 3.0 with higher values be better, i.e. lower levels of depression.
Time Frame: Post-post survey: One year after the intervention
Population: Children ages 10-12 from three tribal communities that included children with their family caregiver who were recruited in schools. Children who responded were recruited into program group. Children who did not respond to participate in the program were allocated to comparison group. Some children did not have valid depression scale data.
Measure: Mean (95% Confidence Interval); unit: change in units on scale
Arm/Group | Program Group | Comparison Group
Number analyzed (Participants) | 137 | 127
change in units on scale | 0.06 [0.01 to 0.11] | -0.01 [-0.07 to 0.05]
Statistical Analysis 1: Comparison: Program Group vs Comparison Group; Test type: Superiority; p = .075, Mixed Models Analysis; Mean Difference (Final Values) = .07, 95% CI 2-sided [-.01 to 0.15]

ADVERSE EVENTS:
Time Frame: 2014-2019. This was a five-year study. with each child participant followed over one year, and during this one-year time frame, there were no adverse events in any of the communities
Description: Does not differ from clinicaltrials.gov definitions
Groups:
- Program and Comparison Groups: The groups are defined above in previous sections. Intervention children are those who choose to participate with their families in the Family Listening after school intervention. Comparison children are those who are invited but can not participate and therefore are placed in the comparison group to take the pre and post tests.
Arm/Group | Program and Comparison Groups
All-Cause Mortality (participants affected / at risk) | 0/266
Serious Adverse Events (participants affected / at risk) | 0/266
Other Adverse Events (participants affected / at risk) | 0/266

LIMITATIONS AND CAVEATS:
Because of the small number of potential participants in each community, we were not able to analyze statistically changes within each community. Aggregate data analysis however was facilitated because of our long-term partnerships with our tribal research teams in each community.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03142009/Prot_SAP_000.pdf